CLINICAL TRIAL: NCT04444349
Title: Protective Effect of Coenzyme Q10 Against Negative Inflammatory Response and Organ Dysfunction in Cardiac and Aortic Surgery (PANDA V): a Randomized Controlled Trial
Brief Title: Protective Effect of CoQ10 Against Negative Inflammatory Response and Organ Dysfunction in Cardiovascular Surgery (PANDA V)
Acronym: PANDA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Beijing Anzhen Hospital (Other); West China Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Hong Liu, Investigator of Cardio-Thoracic Surgery, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PANDA V
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cardiovascular Disease
Keywords: inflammatory response
MeSH Terms: conditions — Cardiovascular Diseases | interventions — coenzyme Q10; Ubiquinone

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coenzyme Q10 group (Experimental): Participants in the experimental group will be given 10mg of Coenzyme Q10 each time (3 times a day).
  Interventions: Drug: Coenzyme Q10
- Control (Sham Comparator): patients only receive standard medical therapy.
  Interventions: Dietary Supplement: Standard Medical Therapy

INTERVENTIONS:
Drug: Coenzyme Q10 — Coenzyme Q10 is a cardiovascular health supplement. It is a component of the electron transport chain and participates in aerobic cellular respiration, which generates energy in the form of ATP. The ingredients in Coenzyme Q10 help regulate the body's production of free radicals, strengthen the arteries and heart, and reverse oxidation.
  Other Names: ubiquinone
  Arms: Coenzyme Q10 group
Dietary Supplement: Standard Medical Therapy — Patients only received standard medical therapy without CoQ10.
  Arms: Control

SUMMARY:
Cardiovascular diseases are the leading causes of death and prescription drug use. Research on certain dietary supplements looks promising as a way to help reduce risk factors. Previous studies showed that CoQ10 levels were decreased in cardiovascular patients and worsening of mitochondrial dysfunction was observed. The overall objective of this study is to determine if supplementing with CoQ10 can reduce inflammatory risk factors in adults with cardiac surgery, independent of other dietary or physical activity changes.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women
* Who receive cardiovascular surgery
* Agree to participate in the surgery and sign the informed consent form

Exclusion Criteria:

* Pregnant or planning on getting pregnant during the study
* Contain a minimum of 2 traits of metabolic syndrome
* Refused to participate in the surgery and refused informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
C-reactive protein | Change from baseline of CRP in mg/L at 5 days after surgery.
  Inflammatory and endothelial blood work biomarkers

SECONDARY OUTCOMES:
Interleukin-6 | Change from baseline of IL-6 in pg/mL at 5 days after surgery.
  Inflammatory and endothelial blood work biomarkers

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No